CLINICAL TRIAL: NCT04291105
Title: Phase 2 Trial of Voyager V1 in Combination With Cemiplimab in Patients With Select Solid Tumors
Brief Title: Phase 2 Trial of Voyager V1 in Combination With Cemiplimab in Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vyriad, Inc. (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VYR-VSV2-203
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Melanoma; Head and Neck Squamous Cell Carcinoma; Colo-rectal Cancer
Keywords: Solid Tumor
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Colonic Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Melanoma intratumoral (Experimental): Melanoma, IT VV1 + IV cemiplimab Patients will receive both treatments on Day 1 and every 3 weeks thereafter until lack of clinical benefit or limiting toxicity. VV1 or cemiplimab can continue after the first dose in combination or as a single agent treatment in subsequent doses.
  Interventions: Biological: VV1; Biological: Cemiplimab
- Head and Neck SCC intratumoral (Experimental): HNSCC, IT VV1 + IV cemiplimab, Patients will receive both treatments on Day 1 and every 3 weeks thereafter until lack of clinical benefit or limiting toxicity. VV1 or cemiplimab can continue after the first dose in combination or as a single agent treatment in subsequent doses.
  Interventions: Biological: VV1; Biological: Cemiplimab
- Colo-rectal Carcinoma intratumoral (Arm closed) (Experimental): (CLOSED) IT VV1 + IV cemiplimab, Patients will receive both treatments on Day 1 and every 3 weeks thereafter until lack of clinical benefit or limiting toxicity. VV1 or cemiplimab can continue after the first dose in combination or as a single agent treatment in subsequent doses.
  Interventions: Biological: VV1; Biological: Cemiplimab

INTERVENTIONS:
Biological: VV1 — VV1 is to be administered on Day 1 and every 3 weeks as long as there is clinical benefit
  Other Names: VSV-IFNβ-NIS, Voyager V1, VV1
Biological: Cemiplimab — Cemiplimab should be given on Day 8 of Cycle 1 (28 days) and then Day 1 of each subsequent 21-day cycle.
  Other Names: Libtayo

SUMMARY:
This is a Phase 2 study designed to determine the preliminary anti-tumor activity and confirm the safety of VV1 in combination with cemiplimab. The study will enroll patients with three distinct separate tumor cohorts. The cancers types are colorectal, head and neck carcinoma, and melanoma that are progressing on CPI treatment.

DETAILED DESCRIPTION:
Patients enrolled into three parallel doublet cohorts with an optimal Simon's two stage design. Patients will receive Voyager V1 as a direct to tumor injection (IT) in all 3 cancer groups and cemiplimab via IV infusion. Patients will return for treatment every 3 weeks until lack of clinical benefit or limiting toxicity. Efficacy evaluations will be conducted every 6 weeks.

ELIGIBILITY:
Inclusion:

1. Age ≥18 years on day of signing informed consent.
2. Specific by tumor cohorts:

   a. For the HSNCC cohort, histologically confirmed diagnosis of advanced and/or metastatic HSNCC suitable for first line immunotherapy.

   i. HPV+ and HPV- patients are allowed.

   ii. Primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx. Participants may not have a primary tumor site of nasopharynx (any histology) or salivary gland tumors.

   iii. PD-L1 status ≥ 1% per local CPS score. Samples should be provided to central lab for post-hoc centralized testing.

   iv. At least 12 months between last dose of prior adjuvant therapy and date of relapse diagnosis (if given). For the purposes of this protocol, "prior adjuvant therapy" only applies to full dose systemic chemotherapy (such as pre-operative systemic induction chemotherapy), but does not include radiation + surgery, or radiation + low or partial dose platinum radiosensitization. There is no time limit (washout) between the end of any prior radiation/ chemoradiation and the start of study drug v. No prior anti-PD-(L)1 treatment for HNSCC.

   b. For the melanoma cohorts, histologically confirmed diagnosis of advanced and/or metastatic cutaneous melanoma for which no existing options are considered to provide clinical benefit.

   i. Best response of uPR, SD or PD to an anti-PD-(L)1-containing regimen.

   ii. Prior anti-PD-(L)1 therapy must have lasted ≥ 12 weeks.

   iii. Radiological progression was demonstrated during or after therapy with a PD-(L)1 immune CPI (only one prior line of PD-(L)1 therapy is permitted.

   iv. If patient received anti-PD-1 as prior adjuvant therapy, patient should have relapsed during therapy or within the subsequent 6 months after last dose. Note: Progression on ipilimumab is not required.

   v. Patients with BRAF V600-positive tumor(s) should have received prior treatment with a BRAF inhibitor (alone or in combination with a MEK inhibitor) in addition to treatment with an anti-PD-1 or to have declined targeted therapy. Note: Patients with BRAF V600-positive tumors with no clinically significant tumor-related symptoms nor evidence of rapidly progressive disease are not required to be treated with a BRAF inhibitor (alone or in combination with a MEK inhibitor) based on investigator's decision

   c. For the CRC cohort, a histologically confirmed diagnosis of advanced and/or metastatic CRC.

   i. Received or are not eligible for standard of care fluoropyrimidine(s), oxaliplatin, irinotecan, anti-VEGF and EGFR-targeted therapies.

   ii. Non-microsatellite instability high (non-MSI high).

   iii. Progression on previous systemic therapy.
3. At least one tumor lesion amenable to IT injection and biopsy that has not been previously irradiated.
4. Measurable disease based on RECIST 1.1., including ≥ 1 measurable lesion(s) to be injected
5. Performance status of 0 or 1 on the ECOG Performance Scale
6. Life expectancy of >3 months.
7. Willingness to provide biological samples required for the duration of the study, including a fresh tumor biopsy sample whilst on study.
8. Adequate organ function assessed by laboratory values obtained ≤14 days prior to enrollment

Exclusion:

Patients meeting any of the following exclusion criteria at screening/Day -1 of first dosing will not be enrolled in the study:

1. Availability of and patient acceptance of an alternative curative therapeutic option.
2. Patients with tumor lesion(s) > 5cm in diameter.
3. Recent or ongoing serious infection, including any active Grade 3 or higher per the NCI CTCAE, v5.0 viral, bacterial, or fungal infection within 2 weeks of registration.
4. Patients who have a diagnosis of ocular, mucosal or acral melanoma.
5. Known seropositivity for and with active infection with HIV.
6. Seropositive for and with evidence of active viral infection with HBV.
7. Seropositive for and with active viral infection with HCV.
8. Known history of active or latent TB.
9. Any concomitant serious health condition, which, in the opinion of the investigator, would place the patient at undue risk from the study, including uncontrolled hypertension and/or diabetes, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease requiring hospitalization within 3 months) or neurological disorder (e.g., seizure disorder active within 3 months).
10. Prior therapy within the following timeframe before the planned start of study treatment as follows:

    1. Small molecule inhibitors, and/or other investigational agent: ≤ 2 weeks or 5 half-lives, whichever is shorter.
    2. Chemotherapy, other monoclonal antibodies, antibody-drug conjugates, or other similar experimental therapies: ≤ 3 weeks or 5 half-lives, whichever is shorter.
    3. Radioimmunoconjugates or other similar experimental therapies ≤ 6 weeks or 5 half-lives, whichever is shorter.
11. NYHA classification III or IV, known symptomatic coronary artery disease, or symptoms of coronary artery disease on systems review, or known cardiac arrhythmias (atrial fibrillation or SVT).
12. Any known or suspected active organ-threatening autoimmune disease, such as inflammatory bowel disease, autoimmune hepatitis, lupus, or pneumonitis, with the exception of hypothyroidism and type 1 diabetes that are controlled with treatment
13. Immunodeficiency or immunosuppression, including systemic corticosteroids at >10 mg/day prednisone or equivalent within 1 week prior to planned start of study treatment.
14. History of Grade 3 or 4 immune-mediated adverse reaction to immune CPIs.
15. Toxicities from previous therapies that have not resolved to a Grade 1 or less.
16. History of non-infectious pneumonitis that required steroids, or current pneumonitis.
17. High volume disease, as assessed clinically by the medical monitor via parameters such as radiologic impression and tumor markers or lactate dehydrogenase (LDH).
18. Portal vein thrombosis involving more than intrahepatic portal vein branches: thrombosis of the right or left portal vein branch or the bifurcation, partial or complete obstruction of the portal vein trunk.

18.19. Known concurrent malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) per imaging assessment | within 24 months
  Percentage of participants with objective response is assessed every six weeks from Cycle 1 Day 1 through disease progression, by investigator review based on RECIST version 1.1

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events assessed by CTCAE v5.0 | within 24 months
  Safety and tolerability
Serum concentration time | within 24 months
  Serum concentration time data using RT-PCR of VSV-IFNβ-NIS and systemic cemiplimab levels
To investigate the pharmacodynamics (PD) of VV1 by measuring serum IFNβ | within 24 months
  To investigate the pharmacodynamics (PD) of VV1 by measuring serum IFNβ expression

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bexon, MD, Study Chair — CMO; Stephen J Russell, MD, Ph.D., Study Director — Clinical Lead
Locations (27):
- United States (23):
  - Mayo Clinical, Phoenix, Arizona
  - City of Hope Medical Center, Durate, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - HOAG Memorial Hospital Presbyterian, Newport Beach, California
  - Saint John's Health Center - John Wayne Cancer Institute (JWCI), Santa Monica, California
  - Stanford Health Care, Stanford, California
  - Yale University, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinical, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Billings Clinic Montana Cancer Consortium, Billings, Montana
  - Atlantic Health, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - UPMC, Pittsburgh, Pennsylvania
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - UT Health San Antonio MD Anderson Cancer Center, San Antonio, Texas
- Brazil (4):
  - Hospital Sao Rafael, Salvador, BR
  - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Amor de Barretos, Barretos, São Paulo

IPD SHARING:
Plan to Share IPD: No